CLINICAL TRIAL: NCT02244736
Title: Changes of the Endothelial Glycocalyx, the Elastic Properties of the Arteries and the Coronary Flow Reserve (CFR) During Oral Glucose Tolerance Test in Patients With New Onset Diabetes Mellitus and First-degree Relatives
Brief Title: Vascular Markers During OGTT in Diabetics and First-degree Relatives
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Assistant Professor in Cardiology, University of Athens
Other Study IDs: K-DM-ATTIKON
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
Keywords: Arterial stiffness; Endothelial glycocalyx; Coronary flow reserve
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Plasma in serum for fibrosis and inflammatory markers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Controls: Subjects with no family history of diabetes mellitus and normal OGTT
- Relatives: First-degree relatives of patients with diabetes mellitus and normal OGTT
- Diabetics: Subjects with abnormal OGTT

SUMMARY:
Arterial stiffness is associated with increased risk for cardiovascular disease. Moreover, the integrity of endothelial glycocalyx plays a vital role in vascular permeability, inflammation and elasticity. The association between damage of endothelial glycocalyx, impaired arterial elastic properties, and CFR in diabetics and first degree relatives has not been explored. The purpose of this study is to explore the association between damage of endothelial glycocalyx, impaired arterial elastic properties, and CFR in diabetics and first-degree relatives before and after during oral glucose tolerance test (OGTT).

DETAILED DESCRIPTION:
The investigators plan to examine 90 subjects without known diabetes a standard 75-gr oral glucose tolerance test (OGTT) will be performed. [30 first degree relatives of diabetics with normal OGTT (relatives), 30 with normal OGTT and no family history of diabetes (normals), and 30 with abnormal OGTT (diabetics) matched for age and sex].

Plasma glucose and serum insulin levels will be measured in venous blood collected at 0, 30, 60, 90 and 120min after glucose loading. At the same time intervals, the investigators will measure:

1. the carotid to femoral pulse wave velocity (PWVc) using the Complior apparatus
2. the aortic pulse wave velocity (PWVa), central systolic blood pressure (cSBP) and augmentation index (AI) using an oscillometric method (Arteriograph,TensioMed) as markers of arterial stiffness and wave reflections
3. the coronary flow reserve (CFR) at baseline and after adenosine infusion (140 μg × kg-1 × min-1) for 3 minutes to assess coronary vasomotor function
4. the perfusion boundary region (PBR- micrometers) of the sublingual arterial microvessels (ranged from 5-25 micrometers) using Sideview Darkfield imaging (Microscan, Glycocheck). Increased PBR is considered an accurate non invasive index of reduced endothelial glycocalyx thickness.

In addition, the investigators will measure free fatty acids, triglycerides, glycerol, C reactive protein (CRP), transforming growth factor-b (TGF-b), Lipoprotein-Associated Phospholipase A2, (LP-LPA2), tumor necrosis factor (TNF-a), interleukin 6 (IL6) and interleukin 10 (IL10) propeptide of type I procollagen, (PIP), propeptide of procollagen type III (PIIINP), matrix metallopeptidases 9 and 2 (MMP 9 and 2), macrophage-colony stimulating factor ( MCSF).

The investigators will measure insulin resistance a) after fasting, using homeostatic model assessment (HOMA) and hepatic insulin sensitivity (HIS) b) during oral glucose tolerance test (OGTT) using Matsuda index and insulin sensitivity index (ISI). The investigators will categorize patients in those with normal (<140 mg/dl at 120 min) and those with abnormal OGTT (>200mg/dl at 120min).

ELIGIBILITY:
Inclusion Criteria:

* subjects without known diabetes
* first degree relatives of diabetics

Exclusion Criteria:

* coronary or valvular heart disease
* congestive heart failure
* peripheral vascular disease
* liver or kidney failure
* history of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 90 subjects, 30 first degree relatives of diabetics withnormal OGTT (relatives), 30 withnormal OGTT and no family history of diabetes (normals), and 30 with abnormal OGTT (diabetics).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Differences of vascular function at baseline and during OGTT among the 3 groups. | Baseline, 30 min, 60 min, 90 min, and 120 min during OGTT.
  Differences of pulse wave velocity, augmentation index and central aortic blood pressure at baseline and during OGTT among the 3 groups.
Differences of endothelial function at baseline and during OGTT among the 3 groups. | Baseline, 30 min, 60 min, 90 min, and 120 min during OGTT.
  Differences of coronary flow reserve and endothelial glycocalyx thickness at baseline and during OGTT among the 3 groups.

SECONDARY OUTCOMES:
Insulin resistance and arterial stiffness | Baseline, 30 min, 60 min, 90 min, and 120 min during OGTT.
  Association of insulin resistance with changes of pulse wave velocity, augmentation index and central aortic blood pressure during OGTT
Insulin resistance and endothelial function | Baseline, 30 min, 60 min, 90 min,120 min of OGTT
  Association of insulin resistance with changes of coronary flow reserve and endothelial glycocalyx during OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; George Pavlidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Vaia Lambadiari, MD, Principal Investigator — 2nd Department of Internal Medicine , University of Athens, Greece; Charalambos Koukoulis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Fotini Kousathana, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; Maria Varoudi, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Vlasios Tritakis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Helen Triantafyllidi, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; George Dimitriadis, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; John Lekakis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece
Locations (1):
- ''Attikon'' University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Ikonomidis I, Lambadiari V, Pavlidis G, Koukoulis C, Kousathana F, Varoudi M, Spanoudi F, Maratou E, Parissis J, Triantafyllidi H, Paraskevaidis I, Dimitriadis G, Lekakis J. Insulin resistance and acute glucose changes determine arterial elastic properties and coronary flow reserve in dysglycaemic and first-degree relatives of diabetic patients. Atherosclerosis. 2015 Aug;241(2):455-62. doi: 10.1016/j.atherosclerosis.2015.06.006. Epub 2015 Jun 9. PMID 26081121